CLINICAL TRIAL: NCT01017718
Title: Prevalence of Pathological Nerve Conduction Velocity in Children and Adolescents Suffering From Diabetes Mellitus Type I
Brief Title: Nerve Conduction Velocity in Diabetic Children
Status: Completed | Type: Observational
Sponsor: Landeskrankenhaus Feldkirch (Other)
Responsible Party: Principal Investigator, Burkhard Simma, Simma B, MD, Landeskrankenhaus Feldkirch
Other Study IDs: 01
Record Dates: First submitted 2009-11-20; First posted 2009-11-23 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Diabetes mellitus type I; nerve conduction velocity; Young score; long term vascular complications
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigators intend to study children and adolescents from 8 to 18 years suffering from diabetes mellitus type 1 for more than one year. The patients will undergo a detailed clinical examination for anthropometric data, blood pressure, blood and urine. Motor and sensory nerve conduction velocity will be examined by electrical stimulation using surface patch electrodes. The nerves to be examined are the nervus tibialis anterior, nervus medianus and nervus peroneus.

Primary outcome:

How many children and adolescents suffering from diabetes mellitus type 1 (duration of disease > 1 year, age 8 to 18a, insulin requirement > 0.5 IU/kg/d) show pathological nerve conduction velocity?

Secondary outcome:

Is there a significant difference in nerve conduction velocity between the group of diabetic patients and the control group of healthy young people? Does the quality of disease control have an influence on nerve conduction velocity? Is there a correlation between nerve conduction velocity in our study patients and the Young Score? Is there a correlation between pathological nerve conduction velocity and other long-term vascular complications (nephropathy, retinopathy)?

DETAILED DESCRIPTION:
Diabetes mellitus type 1 is a chronic disease in which the pancreas no longer produces enough insulin and the glucose in the blood cannot be absorbed into the cells of the body. The main symptom is hyperglycemia. After 10 to 15 years of disease long-term vascular complications including retinopathy, nephropathy, neuropathy, and macrovascular disease are seen. Among the most common long-term complications of diabetes, diabetic neuropathy (DN) is a significant source of morbidity and mortality. There is considerable uncertainty about the prevalence of DN due to a lack of large epidemiological studies and consensus on diagnostic criteria with data variation ranging from 5% to 100%. DN is thought to result from diabetic microvascular injury involving small blood vessels that supply nerves (vasa nervorum). It is a set of heterogeneous clinical syndromes that affect distinct regions of the nervous system, individually or combined. The investigators differentiate autonomic and peripheral neuropathy: Clinical presentation of autonomic neuropathy includes postural hypotension, vomiting, diarrhea, bladder paresis, impotence, sweating abnormalities, and gastric fullness. Peripheral neuropathy presents as altered pain sensations (dys-, para-, hypo- or hyperesthesia), burning, and either superficial or deep pain. The examination of choice for the diagnosis of peripheral neuropathy is to determine nerve conduction velocity.

One of the main goals in treating children and adolescents suffering from diabetes mellitus type I is to avoid long-term complications by early detection of clinical or, even better, subclinical signs. For this reason, the International Society for Pediatric and Adolescent Diabetes (ISPAD) periodically issues Clinical Practice Consensus Guidelines, particularly for screening for vascular complications. With regard to DN there is still uncertainty about the time frame, intensity and diagnostic method of choice.

The investigators aim to examine children and adolescents from 8 to 18 years suffering from diabetes mellitus type I for more than one year with an insulin requirement of more than 0.5 IU/kg/d. The investigators will exclude children with other chronic diseases, handicapped children or children suffering from cancer or chronic renal impairment, as well as children with other neurological diseases which can also cause a change in nerve conduction velocity, and children with blood glucose levels below 50 or above 350 mg/dl. At the time of the annual check-up the patients will undergo a detailed examination for anthropometric data, blood pressure, blood and urine. Thereafter, motor and sensory nerve conduction velocity will be determined by electrical stimulation using surface patch electrodes. The nerves to be investigated are the nervus tibialis anterior, nervus medianus and nervus peroneus. Finally, the patient will undergo a neurological investigation to calculate his Young Score (Neuropathy Symptom Score).

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents with diabetes mellitus type 1 (duration of disease > 1 year, age 8 to 18a, insulin requirement > 0.5 IU/kg/d)

Exclusion Criteria:

* No consent
* Diabetic children with duration of diabetes < 1 year, age <8 or >18 year or insulin requirement > 0.5 IU/kg/d
* Blood glucose levels <50 or >350 mg/dl
* Children with chronic diseases, handicapped children, children with cancer, chronic renal impairment, or neurological diseases

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children and adolescents with diabetes mellitus type 1 (duration of disease > 1 year, age 8 to 18a, insulin requirement > 0.5 IU/kg/d)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-05; Primary Completion 2010-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
How many children and adolescents suffering from diabetes mellitus type 1 (duration of disease > 1 year, age 8 to 18a, insulin requirement > 0.5 IU/kg/d) show pathological nerve conduction velocity? | One electrophysiological investigation (nerve conduction velocity)

SECONDARY OUTCOMES:
Is there a correlation between nerve conduction velocity in our study patients and the Young Score? | One clinical investigation (Young score)

CONTACTS AND LOCATIONS:
Overall Officials: Burkhard Simma, MD, Prof, Principal Investigator — Landeskrankenhaus Feldkirch
Locations (1):
- Department of Pediatrics, University Teaching Hospital, Landeskrankenhaus Feldkirch, Feldkirch, Austria

REFERENCES:
- [Background] Trotta D, Verrotti A, Salladini C, Chiarelli F. Diabetic neuropathy in children and adolescents. Pediatr Diabetes. 2004 Mar;5(1):44-57. doi: 10.1111/j.1399-543X.2004.00041.x. PMID 15043690
- [Background] dos Santos LH, Bruck I, Antoniuk SA, Sandrini R. Evaluation of sensorimotor polyneuropathy in children and adolescents with type I diabetes: associations with microalbuminuria and retinopathy. Pediatr Diabetes. 2002 Jun;3(2):101-8. doi: 10.1034/j.1399-5448.2002.30207.x. PMID 15016164
- [Background] Nelson D, Mah JK, Adams C, Hui S, Crawford S, Darwish H, Stephure D, Pacaud D. Comparison of conventional and non-invasive techniques for the early identification of diabetic neuropathy in children and adolescents with type 1 diabetes. Pediatr Diabetes. 2006 Dec;7(6):305-10. doi: 10.1111/j.1399-5448.2006.00208.x. PMID 17212597
- [Background] Meh D, Denislic M. Subclinical neuropathy in type I diabetic children. Electroencephalogr Clin Neurophysiol. 1998 Jun;109(3):274-80. doi: 10.1016/s0924-980x(98)00017-4. PMID 9741795
- [Background] Hyllienmark L, Brismar T, Ludvigsson J. Subclinical nerve dysfunction in children and adolescents with IDDM. Diabetologia. 1995 Jun;38(6):685-92. doi: 10.1007/BF00401840. PMID 7672490
- [Background] Dorchy H, Noel P, Kruger M, de Maertelaer V, Dupont E, Toussaint D, Pelc S. Peroneal motor nerve conduction velocity in diabetic children and adolescents. Relationships to metabolic control, HLA-DR antigens, retinopathy, and EEG. Eur J Pediatr. 1985 Nov;144(4):310-5. doi: 10.1007/BF00441770. PMID 3865772